CLINICAL TRIAL: NCT00444704
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PRA-027 Administered Orally to Healthy Japanese Females
Brief Title: Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PRA-027 Administered to Healthy Japanese Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3208A1-1002
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Uterine Leiomyomata (Fibroids)
MeSH Terms: conditions — Myofibroma; Leiomyoma

INTERVENTIONS:
Drug: PRA-027

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of ascending single oral doses of PRA-027 in healthy Japanese females. The secondary purpose is to provide the initial pharmacokinetic and pharmacodynamic profiles of PRA-027 in healthy Japanese female subjects.

ELIGIBILITY:
INCLUSION CRITERIA

1. Women of nonchildbearing potential aged 20 to 64 years. Must have a negative pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound scan.
2. Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight must be at least 45 kg.
3. Healthy as determined by the investigator on the basis of screening evaluation.

EXCLUSION CRITERIA

1. Any significant cardiovascular, hepatic, renal, respiratory, gynecologic gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
2. Any history of drug abuse or admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements.
3. Use of any investigational drug within 90 days before study day 1, use of any prescription drug within 30 days before study day 1, consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or cola) or alcoholic beverages within 48 hours before study day 1, consumption of grapefruit or grapefruit-containing products within 72 hours before study day 1, use of any over-the-counter drugs, including herbal supplements (except for the occasional use of vitamins ≤100% of the recommended daily allowance), within 14 days before study day 1, or the donation of blood within 90 days before study day 1.

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-03; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to asess the safety and tolerability of ascending single oral doses of PRA-027 in healthy Japanese females.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tsukuba, Ibaraki, Japan